CLINICAL TRIAL: NCT01263418
Title: A Phase II Trial Of Ofatumumab In Older (≥70 Years) Patients With Previously Untreated Low Or Intermediate Risk Indolent B-Cell Lymphomas
Brief Title: Ofatumumab In Older Patients With Untreated Low Or Intermediate Risk Indolent B-Cell Lymphomas
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients enrolled and funding has been withdrawn.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1018; IRB # 10-1910 (Other: Office of Human Research Ethics)
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Low-Grade; Lymphoma, Intermediate-Grade
Keywords: Follicular Lymphoma; Marginal Zone Lymphoma; Non-Hodgkins Lymphoma; Elderly; Newly Diagnosed; Lineberger Comprehensive Cancer Center; University of North Carolina; Ofatumumab; Arzerra; Phase 2; Geriatric; Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ofatumumab (Experimental)
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — Intravenous; Dosage: 1000mg; Frequency: one time per week; Duration: 8 weeks
  Other Names: ARZERRA; (BLA) 125326

SUMMARY:
This research study will only include two types of non-Hodgkin Lymphoma (NHL), follicular lymphoma or marginal zone lymphoma and participants will be age 70 or older.

The purpose of this research study is to learn about the safety of the treatment with the drug ofatumumab to find out what effects, both good and bad this treatment has on lymphoma. Ofatumumab is a monoclonal antibody. Monoclonal antibodies are being used to treat some types of cancer. Monoclonal antibodies are a type of protein made in a laboratory that can bind substances in the body including cancer cells. Ofatumumab binds to the protein called CD20, which is found on B-cells and lymphoma cells.

The study drug, Ofatumumab, is approved by the United States Food and Drug Administration (FDA) for treatment of other types of blood cancer and is not approved for use in patients with non-Hodgkin Lymphoma. The use of ofatumumab in this study is considered investigational.

In addition to learning about ofatumumab, the researchers are interested in learning about how this cancer treatment affects daily activities. Participants will be asked to complete a Geriatric Assessment (GA). GAs are designed to gather information on memory, nutritional status, mental health, and level of social support. This assessment will help the health care team understand a participant's "functional age" as compared to a participant's actual age.

The researchers also want to collect blood samples to study molecules in follicular lymphoma cells called 'biomarkers' to learn about how the lymphoma responds to therapy. A biomarker is a molecule (for example, DNA or protein) found in the blood or tissues that is a marker for disease. In this study, the investigators will measure the changes of the biomarker called bcl-2. This biomarker research will only be in subjects with follicular lymphoma.

DETAILED DESCRIPTION:
This multicenter Phase II clinical study will investigate the overall response rate (ORR) after 2 months of therapy with weekly ofatumumab in older (≥70 years of age) patients with previously untreated low or intermediate risk indolent NHL (n=37). Secondary objectives include progression free survival (PFS) at 2 years, and an evaluation of the toxicity and tolerability of ofatumumab in this population.

We will also evaluate molecular response to ofatumumab by performing PCR analysis for BCL2/IgH from the peripheral blood.

We will conduct an exploratory analysis of the minimum observed serum concentration (Cmin) of ofatumumab prior to the last dose and correlate this level with ORR.

This trial includes administration of a Geriatric Assessment (GA) tool which patients will be asked to complete serially during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Stage II, III, or IV follicular or marginal zone B-cell CD20+ lymphomas not previously treated with systemic therapy
* Low/intermediate risk grade 1 or 2 follicular NHL or marginal zone lymphoma defined by 2004 Follicular Lymphoma International Prognostic Index (FLIPI) scores
* Measurable disease as assessed by 2 dimensional measurement by CT and/or by bone marrow histopathology.
* Age ≥ 70 years at time of informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy of at least 3 months
* Documented negative serologic testing for human immunodeficiency virus (HIV)
* Documented negative serologic testing for Hepatitis B (HB); this is defined as negative for HBsAg;
* If negative for HBsAg but HBcAb positive (regardless of HBsAb status), an hepatitis B virus (HBV) DNA test will be performed and must be negative for eligibility. Those with negative HBV DNA may be included but must undergo HBV DNA PCR testing every 2 months (see Time and Events table). Prophylactic antiviral therapy may be initiated at the discretion of the investigator in these patients.
* Adequate bone marrow function (without transfusion support within four weeks of screening) as demonstrated by:

  * Hemoglobin ≥ 8 g/dL
  * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
  * Platelet count ≥ 50,000/mm3
* Adequate hepatic and renal function as demonstrated by:

  * Aspartate aminotransferase (AST/ALT) ≤ 2.5 × upper limit of normal (ULN)
  * Total serum bilirubin ≤ 1.5 × ULN
  * Alkaline phosphatase ≤ 2.5 × ULN
  * Serum creatinine ≤ 1.5 × ULN
* If sexually active male with female partner of reproductive capability, has agreed to use a medically accepted form of contraception from time of enrollment to completion of initial follow-up study visit. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method, or total abstinence.
* Signed an institutional review board (IRB)-approved informed consent document for this protocol

Exclusion Criteria:

* Prior therapies for lymphoma except involved field radiation therapy
* Prior anti-CD20 monoclonal antibody or alemtuzumab within 3 months prior to first infusion of ofatumumab for any reason
* Evidence of transformation to aggressive lymphoma
* More than 10 x 109/L circulating CD20+ lymphoma cells
* History of previous allergic reactions to compounds of similar biological or chemical composition as ofatumumab
* Medical or other condition that would represent an inappropriate risk to the patient or would likely compromise achievement of the primary study objective
* Other past or current malignancies with the exception of:

  * Patients who have been free of malignancy for at least 5 years
  * Completely resected, non-melanoma skin cancer
  * Successfully treated in situ carcinoma
* Patients who have current active hepatic or biliary disease (with exception Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to first infusion of ofatumumab, whichever is longer, or currently participating in any other interventional clinical study
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C.
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to first infusion of ofatumumab, congestive heart failure (NYHA III-IV), and arrhythmia (unless controlled by therapy), with the exception of extra systoles or minor conduction abnormalities.
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HBV DNA test will be performed and if positive the patient will be excluded.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2016-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
To determine overall response rates (ORR) following ofatumumab treatment in older (≥ 70 years old) patients with previously untreated low or intermediate risk indolent NHL | 2 years
  The ORR will be evaluated as the rate of complete responses (CR) + partial responses (PR) as defined by the Revised Response Criteria for Malignant Lymphoma (RRCML)

SECONDARY OUTCOMES:
To determine the complete response rate (CR) following ofatumumab treatment in older patients without prior systemic therapy for low or intermediate risk indolent NHL | 2 years
To evaluate the toxicity and tolerability of ofatumumab treatment in the study population | 2 years
Estimate progression free survival (PFS) at 2 years after ofatumumab treatment | 4 years
  PFS is defined as the time from study entry until lymphoma progression or death as a result of any cause.
Evaluate molecular response to ofatumumab therapy by performing PCR analysis for BCL2/IgH from the peripheral blood at baseline and 3 months from initiation of treatment | 3 years
  Molecular response is defined as the percentage of patients with detectable BCL2 PCR at baseline who convert from BCL2 PCR-detectable to undetectable disease status in the peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Park, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center website — http://unclineberger.org/